CLINICAL TRIAL: NCT05054556
Title: Prognostic Value of Galectin-3 for Success of Respiratory Weaning
Brief Title: Galectin and Respiratory Weaning
Acronym: Gal-3
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Asklepios Neurological Clinic Bad Salzhausen (Other)
Collaborators: Asklepios Schlossberg Clinic Bad Koenig (Unknown)
Responsible Party: Sponsor
Other Study IDs: Galectin14092021
Record Dates: First submitted 2021-09-14; First posted 2021-09-23 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-06

CONDITIONS: Galectin-3 During Respiratory Weaning

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Labaratory tests — Estimation of serum levels of the following parameters:
  galectin-3, proBNP, TNI, proGRP, CA15-3, CK, creatinine, urea, crp, pct, leucozytes

SUMMARY:
Galectin-3 is a biomarker for fibrotic activity. In the course of invasive ventilation, fibrotic changes in the lungs may occur. The study aims to investigate whether the level of galectin-3 levels correlates with clinical weaning parameters.

DETAILED DESCRIPTION:
Galectin-3 (Gal-3) is a protein with an important role in cell-cell adhesion, cell-matrix interactions, macrophage activation, angiogenesis, metastasis and apoptosis. Galectin-3 is expressed in the nucleus, cytoplasm, mitochondrion, cell surface, and extracellular space.It is involved in different biological processes: cell adhesion, cell activation and chemoattraction, cell growth and differentiation, cell cycle, and apoptosis. Several studies revealed the function of galectin-3 in cancer, inflammation and (lung) fibrosis, heart disease, and stroke. Expression of galectin-3 is associated with heart failure, including myofibroblast proliferation, fibrogenesis, tissue repair, inflammation, and ventricular remodeling. A correlation between galectin-3 expression levels and various types of fibrosis has been found. Galectin-3 is upregulated in idiopathic pulmonary fibrosis.

Mechanical ventilation can cause lung damage, or worsen it if already present. This phenomenon is called ventilation-induced lung damage. Main mechanisms are high tidal volumes causing overexpansion of the lungs (volutrauma), high airway pressure (barotrauma) and cyclical collapse and reopening of atelectatic alveolar regions (atelectrauma) leading to a pulmonary inflammatory reaction called "bio-trauma".

To evaluate the (potential) lung injury serum levels of galectin-3 are measured on admission to our hospital. During respiratory weaning invasiveness of ventilation will be reduced. Data relating biomarkers especially galectin3 during/after successful respiratory weaning are missing.

This is why follow up measurements of galectin-3 will be done and correlated with ventilation parameters/duration/ success of respiratory weaning.

Prior studies evaluated the role of proGRP and CA 15-3 in patients with lung fibrosis. As a part of the study galectin-3 serum levels will be correlated with serum levels of proGRP and CA 15-3.

In summary the aim of this study is to evaluate the diagnostic value of galectin-3 in respiratory weaning.

ELIGIBILITY:
Inclusion Criteria:

* written informed consent
* mechanical ventilation

Exclusion Criteria:

* history of pulmonary disease
* left ventricular ejection fraction<45%
* missing declaration of consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with mechanical ventilation who are admitted to our hospital for respiratory weaning.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
To correlate the serum levels of galectin-3 and duration of respiratory weaning. | 2-3 months
  Labaratory test+Clinical data.

SECONDARY OUTCOMES:
Serum levels of galectin-3 on admission, after weaning and discharge from hospital. Correlation of: galectin-3 and duration of respiratory weaning invasiveness of ventilation parameters and galectin-3 serum levels of galectin-3, proGRP and CA 15-3. | 2-3 months
  Clinical data, labaratory tests.

CONTACTS AND LOCATIONS:
Locations (2):
- Germany (2):
  - Asklepios Schlossberg Klinik Bad König, Bad König
  - Neurologische Klinik Bad Salzhausen, Nidda

IPD SHARING:
Plan to Share IPD: No